CLINICAL TRIAL: NCT03296631
Title: Phages Dynamics and Influences During Human Gut Microbiome Establishment
Acronym: METAKIDS
Status: Terminated | Type: Observational
Why Stopped: The Pi has estimated that he has received sufficiently biological samples and associated data. it's no longer worth following up.
Sponsor: Institut Pasteur (Industry)
Collaborators: City of Orsay (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2016-097; ID RCB number : 2017-A00750-53 (Other: French national registration number of the study)
Record Dates: First submitted 2017-08-01; First posted 2017-09-28 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Human Gut Microbiome Development
Keywords: microbiome; gut; infant gut; phages; phages-bacteria interactions; microbiome development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fresh stools in diapers. Genomic DNA will be extracted from feces but no human genetic analysis will be realized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children: Enrollment of 15 to 20 children (< 9 months old) at the early beginning of their entry in nursery (crèche) between August and November 2017.
  This cohort will be followed during a maximum period of 36 months . Diapers with fresh stools will be collected once a week per child and then frozen.
  Spontaneous personal day care informations given by the parents to the nurses and recorded in each child's daily logbook will be collected for the research. No specific interviews will be conducted.
  Interventions: Other: collection of diapers with fresh stools

INTERVENTIONS:
Other: collection of diapers with fresh stools — collection of diapers with fresh stools

SUMMARY:
Microbial communities are key components of human environment. Consequently, human gut microbiome have been extensively studied providing a better understanding of the relations between bacterial populations and host physiology. However, a typical analysis tends to elude the complexity of the mixes in term of species, strains, as well as extra-chromosomal DNA molecules such as and phages. MetaKids project aims at bringing, at an unprecedented resolution, a new view of those populations and the internal relationships during human gut establishment, a crucial step with long-term impacts on host health. This project relies on the ability of Meta3C, a newly technique developed in the lab, to identify the bacterial host genomes of the different phages the investigators will detect thanks to the physical collision these molecules experience. Given the role that human gut phages may play in shaping the development of host microbiomes, their potential for application is of great interest.

DETAILED DESCRIPTION:
Over the last decade, the role of microorganisms residing in human intestines has been intensively studied. The intestinal microbiome includes bacteria, viruses, fungi and archaea. The importance of microbiome to human health is highlighted by the observation that dysbiotic shifts in these microbial communities have been associated with numerous human diseases, including obesity, inflammatory bowel disorders, autoimmune disease or gastrointestinal cancer. It is also clearly established that some of these microorganisms interact with the immune system and contribute to its development. The intestinal microbiome is established soon after birth, and its composition changes over the next several years toward a stereotypical 'adult-like' bacterial community structure. Epidemiological studies have demonstrated the importance of this period for a long-term health. It also has been shown that this process can be influenced by multiple interacting factors such as nutrition, antibiotic use and others environmental factors. Much less is known on the viral part of human microbiome. Most of them are phages (phageome) that are known to modulate microbial population through predation or transfer of genetic information between bacteria, and are likely to have important effects on intestinal microbiome establishment and, consequently, human physiology. MetaKids project aims at understanding how the gut phageome develops during the early human life and how it influences the composition of the bacterial microbiome. The investigators will carry a longitudinal study of 15-20 infants from 3-9 months till age 24-30 months. By combining latest metagenomic methods, will be investigated: 1) the composition, evolution and dynamic of the phageome and bacterial microbiome over this critical period; 2) the interactions between phages and bacteria and their relationships; and 3) the impact of environmental factors, like vaccinations or antibiotics treatment on the phages populations. The project is based on the combination of innovative recent metagenomic techniques developed in the lab. DNA is an ubiquitous and stable molecule that can be used as a marker of "compartmentalization" at cellular and population levels, providing important information regarding the genomic structure of a mix of species. Therefore, by combining approaches like purification of virales particles and 3C related methods, the investigators propose to characterize infant gut microbiome establishment and decipher the relationships between the different genomic entities present during this period. This project will bring crucial data on the role of phages during early life of human intestinal tract. Intervention to modify/control intestinal population is a dynamic field and MetaKids project will bring new perspectives for this research area.

ELIGIBILITY:
Inclusion Criteria:

1. Child attending at least 4 days a week one of the two municipal municipal nursery (crèches) in the town of Orsay (91, France);
2. Aged less than 9 months at the time of entry to the crèche (August-October 2017);
3. Parent (s) / legal representative not opposed to the child's participation in the research;

Exclusion Criteria:

* Toilet training;
* Prematurity;
* Participation in clinical research requiring the use of a drug.

Ages: 10 Weeks to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children being in age to attend in a nursery day care structure of the town of Orsay (France) and aged less than 9 months.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Characterization of phages and bacteria genomes during infant gut development. | 3 years
  Genomic reconstruction and characterization of the different genomes (phages, bacteria, yeast) present in the human gut during the three first years of life. This outcomes will provide a large catalog of DNA sequences.
Characterization of phages and bacteria abundance and variations during infant gut development | 3 years
  Characterization of the variation of the different species present in human gut during the 3 first years of life. This outcomes will provide access to the dynamics of the different species present during this period and possibility to correlate them with environmental variation (dietary, age)
Characterization of phages-bacteria interactions | 3 years
  Phages are the major predator of bacteria but their role during human gut establishment remains poorly characterized. This catalog of interactions will allow to understand the role of the phages during human gut development

SECONDARY OUTCOMES:
Characterization of phages and bacteria variations in response to environmental perturbations during infant gut development | 2 to 3 weeks
  Characterization of the small variations of the different species present in human gut during the 3 first years of life in response to environmental perturbations. This outcome will provide access to the dynamics of the different species present during this period and possibility to correlate them with environmental perturbations (antibiotic, vaccine, illness).

CONTACTS AND LOCATIONS:
Overall Officials: Martial Marbouty, Study Director — Institut Pasteur / CNRS
Locations (2):
- France (2):
  - Crèche du Parc, Orsay, Essonne
  - Crèche La Farandole, Orsay, Essonne

IPD SHARING:
Plan to Share IPD: No